CLINICAL TRIAL: NCT03322488
Title: Local Installation of Acetylcysteine, Doxycycline and Fibrin Glue and Surgical Closure of Fistula Openings for Treatment of Perianal Fistulae. An Open Label, Prospective, Multicentric Pilot Study
Brief Title: Fistulodesis Pilot Study for Closure of Perianal Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2016-01310
Record Dates: First submitted 2017-07-10; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Perianal Fistula; Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Doxycycline; Metronidazole; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: 20 patients with Crohn's disease and 20 patients without Crohn's disease will be recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Crohn's Disease (Experimental): 20 patients with Crohn's Disease. Intervention: Fistulodesis
  Interventions: Procedure: Fistulodesis
- Patients without IBD (Experimental): 20 patients without underlying Inflammatory Bowel Disease. Intervention: Fistulodesis
  Interventions: Procedure: Fistulodesis

INTERVENTIONS:
Procedure: Fistulodesis — Fistulodesis comprises the following treatment steps:
  * Curettage and/or brushing of the fistula tract
  * Mini-excision of the inner (endoanal) fistula opening
  * Flushing of fistula tract with acetylcysteine (Concentration: 100mg/ml, max. dosage: 20ml)
  * Flushing/ filling of fistula tract with doxycycline (Concentration: 20mg/ml, max. dosage: 10ml)
  * Filling the fistula tract with fibrin-glue (Evicel®). The maximum amount of Evicel® injected will be 20 ml of the combined product.
  * Surgical closure of inner (endoanal) fistula opening using a Z-suture (Vicryl 3.0)
  * Surgical closure of the outer fistula opening using a Z-suture (Vicryl 3.0)
  Metronidazole and ciprofloxacin will be used at 500mg two times per day for 10 days after the intervention (baseline).
  Other Names: Acetylcystein; Doxycycline; Evicel®; Metronidazole; Ciprofloxacin

SUMMARY:
In this pilot study a new surgical treatment approach for perianal fistulae, called Fistulodesis, is performed. The study aims to assess effectiveness, safety and tolerability of the Fistulodesis procedure. The investigators are aiming to include 20 patients with Crohn's disease and 20 patients without underlying Crohn's disease. It is an open label study with an anticipated duration from January 2017 to January 2020.

DETAILED DESCRIPTION:
The investigators want to test Fistulodesis as a new treatment option which combines established low-invasive surgical and medical treatment steps with the local application of acetylcysteine, doxycycline and fibrin glue in the fistula tract.

Fistulodesis comprises the following steps:

* Curettage of fistula tract
* Mini-excision of the inner (endoanal) fistula opening
* Flushing of fistula tract with acetylcysteine
* Flushing/ filling of the fistula tract with doxycycline
* Filling the fistula tract with fibrin glue
* Surgical closure of inner (rectal) and outer (skin) fistula openings with a Z-suture
* Antibiotic treatment with metronidazole/ ciprofloxacin for 10 days after surgery

Agglutination of the fistula tract is a central part of this study. Agglutinative properties of doxycycline are frequently used by pneumologists for pleurodesis (artificial adhesion of the pleurae to occlude the pleural space for the treatment of pneumothorax or other conditions). Doxycycline (or tetracycline) is thereby instilled into the pleural space, leading to local inflammation and finally pleurodesis. Pleurodesis is an efficient procedure with closure rates >80%. The investigators are expecting to achieve high closure rates also for fistulae.

ELIGIBILITY:
Inclusion Criteria:

* All patients:

  * Signed informed consent
  * Male or female patients ≥18 years of age
  * Perianal fistula existing for at least 3 months
  * Perianal fistula that requires an examination under anaesthesia (EUA)
  * Women of childbearing potential must agree to use effective contraception (for details see chapter 8.6) for the duration of the trial
  * Women of childbearing potential: A negative pregnancy test before inclusion into the trial is required
  * Simple fistula, the whole fistula system must be accessible by curettage or brushing
* Crohn's disease (CD) patients only:

  * CD diagnosis established for ≥3 months
  * CD in remission (Harvey-Bradshaw Index ≤4)

Exclusion Criteria:

* All patients:

  * More than 2 external fistula openings
  * History of irradiation of the anorectum
  * Acute perianal abscess.
  * Perianal operation during the last 4 weeks.
  * Known allergy or non-tolerance against either acetylcysteine, doxycycline, Evicel®, metronidazole or ciprofloxacin.
  * Current antibiotic therapy
  * Severe uncontrolled additional medical, surgical or psychiatric condition, requiring active management
  * Current enrollment into a clinical trial interfering with the endpoints or enrollment in another study for treatment of perianal fistula during the last 4 weeks
  * Inability to follow the procedures of the study, e.g. due to language problems, psychiatrical disorders, dementia, etc. of the participant,
  * Previous enrollment into the current study
  * Women who are pregnant or breastfeeding
  * Intention to become pregnant during the course of the study
  * Large pocket (≥ 1cm) within fistula tract
  * Horseshoe shape of the fistula tract
  * Superficial fistula according to clinical examination and/or ultrasound: (Male patients: Fistula tract involves less than 30% of anal sphincter apparatus, Female patients: Fistula tract involves less than 10% of anal sphincter apparatus)
* Crohn's disease patients only:

  * Evidence of active inflammation in the rectum (besides the fistula)
  * Systemic intake of steroid-medication (currently or during the last 4 weeks) in a dose of >20mg prednisone or equivalent
  * New immunosuppressant medication for Crohn's disease within the last 4 weeks before inclusion into the study (changes in 5-ASA medication or rectal treatment with 5-ASA or budesonide are permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fistulodesis success criteria | week 24
  Closure of all perianal fistula tracts of a patient at week 24 as defined by the presence of all of the following "Fistulodesis success criteria":
  * No secretion from fistula during the last 2 weeks as reported by the patient
  * No secretion upon careful pressing onto fistula tract
  * Fistula tract outer opening macroscopically closed upon inspection
  * No pain at the site of the former fistula opening during gentle pressing

SECONDARY OUTCOMES:
Improvement of quality of life | at week 24
  Improvement of quality of life (IBD-Q) at week 24 compared to baseline
Improvement of PDAI | at week 4, 12, 24
  Improvement of PDAI (Peranal Disease Activity Index) at week 4, 12, 24 compared to baseline
Reduction in fistula activity | at week 4, 12 and 24
  Reduction in fistula activity assessed by fistula drainage assessment (FDA) and "Fistulodesis success criteria" at week 4, 12 and 24 compared to baseline
Risk factors for treatment failure | at week 24
  Risk factors for treatment failure (multivariate analysis)
Comparison of fistula closure rates in patients with CD and patients without IBD | at week 24
  Comparison of fistula closure rates in patients with CD and patients without IBD
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | at weeks 4, 12, 24, 12 months and 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Long-term follow-up | at 12 months and 24 months
  Long-term follow-up (12 months, 24 months after the end of the study): Assessment of the long-term success after 12 and 24 months by telephone. The patients will be asked about possible fistula symptoms (pain, drainage).

OTHER OUTCOMES:
Microbiota composition of fistula tract | material obtained at baseline
  We will analyze the curettage material from the fistula tract by 16S sequencing to determine microbiota composition. We will compare bacterial diversity (number bacterial species) from CD patients and patients without Crohn's disease

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Division of Gastroenterology, University Hospital Zurich, Zurich
  - Bethanien-Klinik, Zurich